CLINICAL TRIAL: NCT02877316
Title: MYPLAN - Effectiveness of a Safety Plan App to Manage Crisis of Persons at Risk of Suicide - a Multi-center, Superiority Randomized Clinical Trial
Brief Title: MYPLAN - Effectiveness of a Safety Plan App to Manage Crisis of Persons at Risk of Suicide
Acronym: MYPLAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Principal Investigator, Kate Aamund, MD, postdoctoral researcher, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MHSCRDenmark
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Suicide Prevention; Suicidal Thoughts; Suicide Attempts
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation; Suicide, Attempted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MYPLAN app (Experimental): MYPLAN app (safety plan) as part of treatment
  Interventions: Other: MYPLAN-safety plan as an application for smart phones
- Safety plan on paper (Active Comparator): Safety plan on paper as part of treatment
  Interventions: Other: safety plan on paper

INTERVENTIONS:
Other: MYPLAN-safety plan as an application for smart phones — MYPLAN app as a integral part of the standard treatment
  Arms: MYPLAN app
Other: safety plan on paper — Standard treatment with safety plan on paper
  Arms: Safety plan on paper

SUMMARY:
Background: Persons with a past episode of self-harm or severe suicidal ideation are at elevated risk of self-harm as well as dying by suicide. It is well established that suicidal ideation fluctuates over time. Safety plans in paper format are mandatory part of the treatment regime in the suicide preventive clinics in Denmark. The aim of the trial is to compare the paper version of the safety plan with a new-developed app in reducing suicide ideation and other symptoms, as an add-on to the supportive psychotherapy delivered in the clinics.

Hypothesis: It is hypothesized that participants randomized to MYPLAN will have lower suicide ideation as well as improvements on the secondary outcomes than users who have the paper version.

Methods: The trial is designed as a 2-arm observer-blinded parallel group randomized clinical superiority trial, where participants will either receive: 1) Experimental intervention: the safety plan provided as the app MYPLAN, or 2) Treatment as Usual: the safety plan in the original paper format. Both intervention groups will also receive standard psychosocial therapeutic care, up to 8-10 sessions of supportive psychotherapy.Based on a power calculation a total of 546 participants, 273 in each arm will be included. They will be recruited from national suicide preventive clinics. Follow-ups will be conducted at 3, 6, 9, and 12 months after date of inclusion.

Participants, inclusion and exclusion criteria: There is no age restriction on participation in the study and all participants will be recruited from the suicide prevention clinics in Denmark. These clinics are highly specialized outpatient care centers, offering short-term supportive psychotherapy and social counselling for suicidal patients. In order to participate in the study, participants must have a smartphone (IPhone or android phone) and understand sufficient Danish to use MYPLAN. Persons having a particularly severe alcohol or substance abuse disorder, which might inflict with skills of orientation and memorywill not be offered participation in the RCT.

Outcomes Patient reported outcomes (PROM) are collected at baseline and follow-up through self-administered tablet/internet-based questionnaires. Primary outcome is suicide ideation. Secondary outcomes are:, hopelessness, depressive symptoms, quality of life, and modified CSQ-8.

Statistical analysis: Data analysis will be based on intention-to-treat principle. We will examine this using repeated measurement in mixed models. Missing data will be handled with multiple imputations.

The trial will start in November 2016 and patient recruitment is expected to finish November 2017. Analysis and results are expected in 2018.

DETAILED DESCRIPTION:
MYPLAN -mobile phone application to manage crisis of persons at risk of suicide:

a multi-center, superiority randomized clinical trial.

Andreasson K, Krogh J, Frandsen H, Buus N, Bech. P Nordentoft M, Erlangsen A Background

In Denmark, there are 8-10,000 people who attempt suicide on a yearly basis1. Suicide ideation is a part of a continuum, where initial suicidal ideation might develop into concrete plans and actions, depending on the suicidal intent suicidal actions might end as suicide attempts or completed suicide2 . Therefore, in order to prevent suicidal behavior and suicides, it is important to avoid or reduce suicide ideation; i.e. securing better control of painful thoughts and the suicidal behavior. This can be done with a safety plan. The safety plan has been developed as a cognitive therapeutic intervention applied empirically in some earlier studies 345. The safety plan can be considered as a part of a cognitive behavior therapeutic intervention, which reduces the suicidal risk and consists of basic components, such as 1) recognizing warning signs of an upcoming suicidal crisis, 2) work with internal coping strategies, 3) distraction from suicidal thoughts, by the use of social contacts and social settings6. This can be done by removing assess of lethal means, and self-monitoring the triggers of the "suicidal mode"7.

To prevent suicidal behavior, The National Board of Health has established Suicide Prevention Clinics nationwide in Denmark. The clinics offering highly specialized short-term supportive psychotherapy and social counselling for suicidal patients in an outpatient setting. The target group is a subsample of all persons with severe suicide ideation or suicide attempts as the clinics focus on persons at risk of suicide who do not have severe underlying psychiatric disorders that required psychiatric admission or specialized treatment8. Some clinics are specialized in children and adolescents and will offer support patients young as 10 years of age. The safety plan is an integral part of the treatment and all patient works with during the first sessions.

Hypothesis The hypothesis of this trial is that an app-based safety plan is more effective than a paper version of a safety plan in reducing suicide ideations in suicidal patients.

Purpose

The purpose of this trial is to investigate if a safety plan delivered as an app compared to a safety plan delivered by paper, can reduce suicide ideation after 12 months intervention in patients referred to Suicide Prevention Clinics.

Methods/design

The trial is designed as a 2-arm, multi-site, parallel group, observer-blinded randomized clinical superiority trial. Based on a power calculation, a total of 546 participants, 273 in each arm will be included, recruited from national suicide preventive clinics. Both groups will receive treatment as usual consisting of short term psychotherapy and social counselling: 1) Experimental intervention the safety plan provided as the app MYPLAN, or 2) Treatment as Usual (TAU): the safety plan in the original paper format.

Recruitment and criteria for inclusion and exclusion

All participants will be recruited through the Suicide Prevention Clinics in Denmark. The patients are referred from somatic and psychiatric wards after suicide attempts, general practitioners, and can also refer themselves to the suicide preventive clinics. There is no age restriction on participation in the study.

Enrollment and randomization

At the first visits at the Suicide Prevention Clinic, eligible participants will receive oral and information about the study as well as an information pamphlet. They will be offered time for reflection and possibility to have renewed appointment at the clinic together with a relative, before answering. If the patient fulfils all the inclusions criteria and none of the exclusion criteria, the patient will be randomized using a computer-generated sequence randomization to either 1) Treatment as usual plus app: treatment as usual plus the safety plan app, or 2) treatment as usual pus safety plan on paper. The randomization will be stratified by gender and previous self-harm (yes/no), and will be facilitated through an external, centrally administered internet service. The clinician working the Suicide Prevention Clinics, will by accessing the internet obtain information on the patients allocation (safety plan either as an app or paper version), immediately after the patients has provided informed consent. This procedure will ensure adequate allocation concealment.

Blinding Due to the nature of the intervention, a blinding of participants and clinicians is not possible, but outcome assessment and analyses will be carried out with blinding of treatment allocation. All data will be collected through questionnaires (SurveyXact) secured on an encrypted server. The analyses will be performed by blinded scientists.

Interventions Treatment as Usual (TAU): Participants allocated to the treatment at usual will receive up to 8-10 sessions of supportive psychotherapy as part of the standard care of the suicide preventive clinics. Each of the clinics apply different or combined therapies including cognitive, problem-solving, crisis, dialectical behavior, integrated care, psychodynamic, systemic, psychoanalytic approaches, and/or social counselling. A uniform treatment algorithm is not followed; elements are chosen on the basis of what is deemed the most promising strategy in each individual case. As an integral part of the therapy the clinical fill in a safety plan with the patient by reviewing what are signs of situations where crises occur and what has previously worked as strategies of distraction as well as help-seeking. The safety plan is presented to the patient using a comparable manual-based instruction. Participants randomized to the paper format will write the safety plan on a sheet of paper and bring home the original while the clinical keeps a copy together with the medical records of the patient.

Experimental intervention: Participants allocated to the experimental intervention will receive the treatment as usual, and have an introduction to the app-based safety plan MYPLAN. Using the instruction manual, the clinician will review previous crisis situations and possible strategies.

See figure 1. CONSORT flow diagram

Outcomes

Primary outcome will be measured as the difference in suicide ideation before entering the trial and after 12 month participation in the trial. This is measured by Becks suicide ideation scale (BSS 21-items). The outcome is considered as a proxy measure for suicide attempt and completed suicide.

Secondary outcomes are: hopelessness (Becks Hopelessness Scale, BHS), depressive symptoms (Major depression Inventory, MDI).

Exploratory outcomes We have chosen some exploratory outcomes such as, quality of life measured by WHO Well-being Index, (WHO-5), user satisfaction will be measured by modified User satisfaction Client Satisfaction Questionnaire (CSQ-8), self-harm (self-reported), mortality, admission to psychiatric or somatic emergency wards, and other somatic and psychiatric hospital registers data.

Patient reported outcomes measures (PROM) These are collected at baseline and follow-up through self-administered tablet-/ internet-based questionnaires. Follow-ups will be conducted at 3, 6, 9, and 12 months after date of inclusion. Participants will receive an e-mail with a link to an online survey. Respondents can log on to a secure data portal, SurveyXact, with their personal trial id-number and answers to questionnaires are collected.

The register-based outcomes such as mortality, suicide attempt, somatic and usage of somatic and mental health care services will be assessed at 12 and 24 months by obtaining data extract from above listed registries.

Statistical analysis

The primary outcome is the mean change in Becks Suicide Ideation scale at 6 months. We expect that participants in the intervention group at 6 months score 2.5 points lower compared to participants in the TAU group. Based on previous publication we expect a post-intervention SD of 9. Setting the alpha level to 5 percent and the beta level to 10 percent we need to include 273 participants for each group to a total of 546 participants.

Analysis of the primary outcome will be conducted according to intention-to-treat principle: all participants will be included in final analysis according to group assignment regardless of adherence to treatment. This study has multiple assessment points and for the primary analysis we will use repeated measurements in a mixed model with unstructured variance. This procedure is able to handle baseline differences and missing data. For participants with missing data in two or more data points we will identify potential differences to participants with full data and use include these variables as potential confounders in secondary analysis.

All statistical analysis will be conducted in SPSS. All tests will be two-tailed and p values below 0.5 will be considered significant and interpreted with respect to hierarchy of hypothesis.

Pilot study/feasibility test

Prior to study being a pilot study will be carried out in one of the sites. The aim is to make the pilot study as similar to the trial as possible. A total of 40 participant will be recruited, 20 in each arm. The randomization and other technical and practical procedures will be tested. Clinicians will present the safety plan as described above using a manual-based instruction. The participants will be followed for 3 months. Data on all scales listed as outcomes will be collected; at the time of enrollment by tablet and at end of follow-up by email.

Ethical considerations The trial will be approved by the Regional Ethics Committee in the Capital Region of Denmark and the Danish Data Protection agency. The trial is registered under Clinicaltrials.gov as NCT. In accordance to with the Consort guidelines, we will publish positive, neutral and negatives findings in the trial. The patients will be informed about the trial both verbally and written information before signing the written consent. They are offered time for consideration and they can have a renew appointment together with a spouse, before signing the written consent. It will be stressed that participation are voluntary. Participation and the written consent can be withdrawn at any time.

Organization and economy The trial is led by postdoctoral researcher Kate Andreasson Aamund, Psychiatric Centre North Zealand in close collaboration with Danish Research Institute for Suicide Prevention (DRIPS), Mental Health Center Copenhagen and the Suicide Prevention Clinics. The patient recruitment will be done through the Danish Suicide Prevention Clinics in Denmark. The project has received funding from the Danish non-profit foundation (TrygFonden).

Analyses and results are expected in summer 2018

ELIGIBILITY:
Inclusion Criteria:

* Smart phone (Iphone/android)
* Understand sufficient Danish to use MYPLAN
* Informed written consent

Exclusion Criteria:

* Alcohol or substance abuse disorder (DSM-V)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 546 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Suicide ideation | 12 month
  Primary outcome will be measured as the difference in suicide ideation before entering the trial and after 6 month participation in the trial. This is measured by Becks suicide ideation scale (BSS 21-items).

SECONDARY OUTCOMES:
Depressiv symptoms | 12 month
  Depressive symptoms measured by Major depression Inventory, MDI)
Hopelessness | 12 month
  Hopelessness measured by Becks Hopelessness Scale, BHS-21items

OTHER OUTCOMES:
Quality of life index | 12 month (Baseline, 3 month,
  Quality of life measured by WHO-5
Satisfaction of the app | 12 month
  Satisfaction measured by a modified version of CSQ-8

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nordentoft, MD, Ph.D MSc, Study Chair — Mental Health Center Copenhagen
Locations (4):
- Denmark (4):
  - Psychiatric centre Ballerup, Clinic for psychoterapy, Ballerup Municipality
  - Competence centre for suicide prevention, Copenhagen
  - Psychiatric Centre North Zealand, Hillerød
  - Clinic for suicide prevention, Køge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Christiansen E, Jensen BF. Register for Suicide Attempts. Dan Med Bull. 2004 Nov;51(4):415-7. PMID 16009065
- [Background] Brown GK, Ten Have T, Henriques GR, Xie SX, Hollander JE, Beck AT. Cognitive therapy for the prevention of suicide attempts: a randomized controlled trial. JAMA. 2005 Aug 3;294(5):563-70. doi: 10.1001/jama.294.5.563. PMID 16077050
- [Background] Stanley B, Brown G, Brent DA, Wells K, Poling K, Curry J, Kennard BD, Wagner A, Cwik MF, Klomek AB, Goldstein T, Vitiello B, Barnett S, Daniel S, Hughes J. Cognitive-behavioral therapy for suicide prevention (CBT-SP): treatment model, feasibility, and acceptability. J Am Acad Child Adolesc Psychiatry. 2009 Oct;48(10):1005-1013. doi: 10.1097/CHI.0b013e3181b5dbfe. PMID 19730273
- [Background] Yanos PT, Stanley BS, Greene CS. Research risk for persons with psychiatric disorders: a decisional framework to meet the ethical challenge. Psychiatr Serv. 2009 Mar;60(3):374-83. doi: 10.1176/ps.2009.60.3.374. PMID 19252051
- [Background] Erlangsen A, Lind BD, Stuart EA, Qin P, Stenager E, Larsen KJ, Wang AG, Hvid M, Nielsen AC, Pedersen CM, Winslov JH, Langhoff C, Muhlmann C, Nordentoft M. Short-term and long-term effects of psychosocial therapy for people after deliberate self-harm: a register-based, nationwide multicentre study using propensity score matching. Lancet Psychiatry. 2015 Jan;2(1):49-58. doi: 10.1016/S2215-0366(14)00083-2. Epub 2015 Jan 8. PMID 26359612
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- [Derived] Andreasson K, Krogh J, Bech P, Frandsen H, Buus N, Stanley B, Kerkhof A, Nordentoft M, Erlangsen A. MYPLAN -mobile phone application to manage crisis of persons at risk of suicide: study protocol for a randomized controlled trial. Trials. 2017 Apr 11;18(1):171. doi: 10.1186/s13063-017-1876-9. PMID 28399909
- See also: Ref. 5. Cognitive therapy for suicidal patients — http://www.apa.org/pubs/books/4317169.aspx
- See also: Ref 7. Why people die by suicide — http://www.hup.harvard.edu/catalog.php?isbn=9780674025493
- See also: Ref. 9. Diagnostic and statistical manual of mental health disorders — https://www.psychiatry.org/psychiatrists/practice/dsm